CLINICAL TRIAL: NCT04024891
Title: Randomized, Cross-Over, Double-Masked, Placebo-Controlled Study of the Safety and Efficacy of Phentolamine Mesylate Ophthalmic Solution to Reverse Pharmacologically Induced Mydriasis in Normal Healthy Subjects
Brief Title: Safety and Efficacy of Ophthalmic Phentolamine Mesylate to Reverse Pharmacologically Induced Mydriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocuphire Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: OPI-NYXRM-201 (MIRA-1)
Record Dates: First submitted 2019-07-11; First posted 2019-07-18 (Actual); Results first posted 2022-08-15 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2022-08

CONDITIONS: Mydriasis; Dilation
Keywords: Nyxol; Pharmacologically Induced Mydriasis; Dilation
MeSH Terms: conditions — Mydriasis; Dilatation, Pathologic

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phentolamine Mesylate Ophthalmic Solution 1% (Experimental): 1 drop in each eye, 1 hour post medically-induced mydriasis
  Interventions: Drug: Phentolamine Mesylate Ophthalmic Solution 1%
- Phentolamine Mesylate Ophthalmic Solution Vehicle (Placebo Comparator): 1 drop in each eye, 1 hour post medically-induced mydriasis
  Interventions: Other: Phentolamine Mesylate Ophthalmic Solution Vehicle (Placebo)

INTERVENTIONS:
Drug: Phentolamine Mesylate Ophthalmic Solution 1% — 1% phentolamine mesylate ophthalmic solution (Nyxol), a non-selective alpha-1 and alpha-2 adrenergic antagonist
  Other Names: Nyxol®; Nyxol
  Arms: Phentolamine Mesylate Ophthalmic Solution 1%
Other: Phentolamine Mesylate Ophthalmic Solution Vehicle (Placebo) — Topical Sterile Ophthalmic Solution
  Arms: Phentolamine Mesylate Ophthalmic Solution Vehicle

SUMMARY:
The objectives of this study are:

* To evaluate the efficacy of Nyxol (phentolamine mesylate ophthalmic solution 1%) to expedite the reversal of pharmacologic mydriasis
* To evaluate the safety of Nyxol
* To evaluate the effect of Lumify® to suppress conjunctival hyperemia (redness) potentially associated with administration of Nyxol

DETAILED DESCRIPTION:
Randomized, 2-arm cross-over, double-masked Phase 2b study in approximately 32 healthy subjects, evaluating safety and efficacy of Nyxol in subjects with pharmacologically induced mydriasis.

At the first visit subjects will be screened for study eligibility.

After screening, eligible subjects will be randomized 1:1 to one of the two treatment sequences:

Treatment sequence 1: Placebo (Visit 1), Nyxol (Visit 2).

Treatment sequence 2: Nyxol (Visit 1), Placebo (Visit 2).

Randomization will be stratified by mydriatic agent (2.5% phenylephrine or 1% tropicamide). Approximately one half of the randomized subjects will receive 2.5% phenylephrine and one half will receive 1% tropicamide. Subjects will receive their mydriatic agent 1 hour before treatment. Each subject will receive the same mydriatic agent throughout the study.

At each visit, pupil diameter (PD), accommodation, near and distance visual acuity (VA) and redness in each eye will be measured before (-1 hour/baseline) and 1 hour after (maximum/0 minutes) the mydriatic agent instillation in each eye (i.e., right before the study treatment is administered), and at 30 minutes, 1 hour, 2 hours, 4 hours and 6 hours after treatment dosing.

As needed, two hours post treatment, subjects may request the administration of Lumify® in the non-study eye.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 and ≤ 45 years of age with brown irides (irises) only
2. Otherwise healthy and well controlled subjects
3. Able to comply with all protocol mandated procedures and to attend all scheduled office visits
4. Willing to give written informed consent to participate in this study

Exclusion Criteria

1. Clinically significant ocular disease as deemed by the Investigator (e.g., cataract, glaucoma, corneal edema, uveitis, severe keratoconjunctivitis sicca) that might interfere with the study
2. Unwilling or unable to discontinue use of contact lenses during treatment visits
3. Ocular trauma, ocular surgery or non-refractive laser treatment within the 6 months prior to screening
4. Ocular medication of any kind within 30 days of screening, with the exception of a) lid scrubs (which may have been used prior to, but not after screening) or b) lubricating drops for dry eye (preservative-free artificial tears), which may be used in between the study treatment days
5. Recent or current evidence of ocular infection or inflammation. Current evidence of clinically significant blepharitis, conjunctivitis, or a history of herpes simplex or herpes zoster keratitis at screening
6. History of diabetic retinopathy
7. Closed or very narrow angles that in the Investigator's opinion are potentially occludable if the subject's pupil is dilated
8. History of any traumatic (surgical or nonsurgical) or non-traumatic condition affecting the pupil or iris (e.g., irregularly shaped pupil, neurogenic pupil disorder, iris atrophy, iridotomy)
9. Known allergy or contraindication to any component of the mydriatic agents or the vehicle formulation
10. Known hypersensitivity or contraindication to α- and/or β-adrenoceptor antagonists (e.g., chronic obstructive pulmonary disease or bronchial asthma; abnormally low blood pressure (BP) or heart rate (HR); second- or third-degree heart blockage or Congestive Heart Failure (CHF); severe diabetes)
11. Clinically significant systemic disease (e.g., uncontrolled diabetes, myasthenia gravis, cancer, hepatic, renal, endocrine or cardiovascular disorders) that might interfere with the study
12. Initiation of treatment with or any changes to the current dosage, drug or regimen of any topical or systemic adrenergic or cholinergic drugs up to 7 days prior to screening, or during the study
13. Participation in any investigational study within 30 days prior to screening
14. Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control. Acceptable methods include the use of at least one of the following: intrauterine device (IUD), hormonal (oral, injection, patch, implant, ring), barrier with spermicide (condom, diaphragm), or abstinence. An adult woman is considered to be of childbearing potential unless she is 1 year postmenopausal or 3 months post-surgical sterilization. All females of childbearing potential must have a negative urine pregnancy test result at Visit 1/Screening and Visit 2 examinations and must intend to not become pregnant during the study
15. Resting heart rate (HR) outside the normal range (50-110 beats per minute) at the Screening Visit. HR may be repeated only once if outside the normal range following at least a 5-minute rest period in the sitting position
16. Hypertension with resting diastolic BP > 105 mmHg or systolic BP > 160 mmHg at the Screening Visit. BP may be repeated only once if outside the specified range following at least a 5-minute rest period in the sitting position

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Kannar Eye Care, Pittsburg, Kansas
  - Kentucky Eye Institute, Lexington, Kentucky
  - Athens Eye Care, Athens, Ohio
  - West Bay Eye Associates, Warwick, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karpecki PM, Foster SA, Montaquila SM, Kannarr SR, Slonim CB, Meyer AR, Sooch MP, Jaber RM, Charizanis K, Yousif JE, Klapman SA, Amin AT, McDonald MB, Horn GD, Lazar ES, Pepose JS. Phentolamine Eye Drops Reverse Pharmacologically Induced Mydriasis in a Randomized Phase 2b Trial. Optom Vis Sci. 2021 Mar 1;98(3):234-242. doi: 10.1097/OPX.0000000000001656. PMID 33633016

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a crossover design study, so all 32 enrolled subjects were included in both treatment groups.
Groups:
- PMOS 1% First, Then PMOS Vehicle: Participant received Phentolamine Mesylate Ophthalmic Solution 1%: 1% phentolamine mesylate ophthalmic solution (Nyxol), a non-selective alpha-1 and alpha-2 adrenergic antagonist at Visit 1. Then, after one week, they received Phentolamine Mesylate Ophthalmic Solution Vehicle (Placebo): Topical Sterile Ophthalmic Solution at Visit 2.
  1 drop in each eye, 1 hour post medically-induced mydriasis at both visits.
- PMOS Vehicle First, Then PMOS 1%: Participants received Phentolamine Mesylate Ophthalmic Solution Vehicle (Placebo): Topical Sterile Ophthalmic Solution at Visit 1. Then, after one week, they received Phentolamine Mesylate Ophthalmic Solution 1%: 1% phentolamine mesylate ophthalmic solution (Nyxol), a non-selective alpha-1 and alpha-2 adrenergic antagonist at Visit 2.
  1 drop in each eye, 1 hour post medically-induced mydriasis for both visits.
Period: Overall Study
Arm/Group | PMOS 1% First, Then PMOS Vehicle | PMOS Vehicle First, Then PMOS 1%
Started | 16 | 16
Completed | 16 | 15
Not Completed | 0 | 1
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Population: Subjects baseline values are included in the column to which they were randomized first in this crossover design trial. One subject in the PMOS Vehicle First, Then PMOS group was found to be pregnant after their first visit and was withdrawn from the trial and did not crossover to receive PMOS, resulting in an analytical sample of n = 31.
Groups:
- PMOS 1% First, Then PMOS Vehicle: 1 drop in each eye, 1 hour post medically-induced mydriasis
  Phentolamine Mesylate Ophthalmic Solution 1%: 1% phentolamine mesylate ophthalmic solution (Nyxol), a non-selective alpha-1 and alpha-2 adrenergic antagonist
- PMOS Vehicle First, Then PMOS 1%: 1 drop in each eye, 1 hour post medically-induced mydriasis
  Phentolamine Mesylate Ophthalmic Solution Vehicle (Placebo): Topical Sterile Ophthalmic Solution
- Total: Total of all reporting groups
Arm/Group | PMOS 1% First, Then PMOS Vehicle | PMOS Vehicle First, Then PMOS 1% | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (8.18) | 28.5 (8.54) | 28.0 (8.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 7 | 5 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Iris Color [Count of Participants; unit: Participants]
  Brown | 16 | 15 | 31
  Non-Brown | 0 | 0 | 0
Mydriatic Agent Recieved [Count of Participants; unit: Participants]
  Phenylephrine | 8 | 7 | 15
  Tropicamide | 8 | 8 | 16
Baseline Pupil Diameter (Study Eye) [Mean (Standard Deviation); unit: mm] | 4.5 (0.80) | 4.5 (0.79) | 4.5 (0.78)
Maximum Dilated Pupil Diameter (Study Eye) [Mean (Standard Deviation); unit: mm] | 7.3 (1.04) | 7.2 (1.04) | 7.3 (1.02)

OUTCOME MEASURES:

1. Primary Outcome: Pupil Diameter (Change From Max)
Description: Change in pharmacologically-induced mydriatic (maximum) pupil diameter at 2 hours post-treatment in the study eye.
Time Frame: 2 hours
Population: Crossover design study
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Phentolamine Mesylate Ophthalmic Solution 1% | Phentolamine Mesylate Ophthalmic Solution Vehicle
Number analyzed (Participants) | 31 | 31
mm | -1.69 (0.117) | -0.69 (0.117)
Statistical Analysis 1: Comparison: Phentolamine Mesylate Ophthalmic Solution 1% vs Phentolamine Mesylate Ophthalmic Solution Vehicle; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -1.0, 95% CI 2-sided [-1.3 to -0.7]

2. Secondary Outcome: Pupil Diameter (Change From Max)
Description: Change in pharmacologically-induced mydriatic (maximum) pupil diameter at remaining timepoints (30 min, 1 hours, 4 hours, 6 hours)
Time Frame: 30 min, 1 hours, 4 hours, 6 hours
Population: Crossover design trial
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Phentolamine Mesylate Ophthalmic Solution 1% | Phentolamine Mesylate Ophthalmic Solution Vehicle
Number analyzed (Participants) | 31 | 31
mm
  30 minutes | -0.06 (0.039) | -0.13 (0.039)
  1 hour | -0.77 (0.072) | -0.29 (0.072)
  4 hours | -2.83 (0.145) | -1.69 (0.146)
  6 hours | -3.24 (0.132) | -2.54 (0.133)

3. Secondary Outcome: Pupil Diameter Return to Baseline
Description: Percent of Subjects Achieving Pupil Diameter No More Than 0.5 mm Above Baseline by Time Point with either phenylephrine or tropicamide
Time Frame: 0 min, 1 hour, 2 hours, 4 hours, 6 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Phentolamine Mesylate Ophthalmic Solution 1% | Phentolamine Mesylate Ophthalmic Solution Vehicle
Number analyzed (Participants) | 31 | 31
Participants
  0 min | 2 | 3
  1 hour | 6 | 3
  2 hour | 11 | 6
  4 hour | 24 | 12
  6 hour | 31 | 28

4. Secondary Outcome: Accommodation Measured by the Near Point Rule (Diopters) (Change From Baseline), Percent With Unchanged Accommodation
Description: Change from baseline (-1 hour) in accommodation at each time point (0 min, 2 hours, 4 hours) with Tropicamide and Phenylephrine
  Worsening of accommodation is defined as an amplitude decrease of greater than 1 diopter compared to baseline
Time Frame: 0 min, 2 hours, 4 hours
Population: Crossover Design Trial
Measure: Count of Participants; unit: Participants
Arm/Group | Phentolamine Mesylate Ophthalmic Solution 1% | Phentolamine Mesylate Ophthalmic Solution Vehicle
Number analyzed (Participants) | 31 | 31
Participants
  Dilated with Tropicamide, 0 min: number analyzed (Participants) | 16 | 16
  Dilated with Tropicamide, 0 min: Unchanged Accommodation | 3 | 2
  Dilated with Tropicamide, 0 min: Changed Accommodation (≥1 D) | 13 | 14
  Dilated with Tropicamide, 2 hr: number analyzed (Participants) | 16 | 16
  Dilated with Tropicamide, 2 hr: Unchanged Accommodation | 7 | 3
  Dilated with Tropicamide, 2 hr: Changed Accommodation (≥1 D) | 9 | 13
  Dilated with Tropicamide, 4 hr: number analyzed (Participants) | 16 | 16
  Dilated with Tropicamide, 4 hr: Unchanged Accommodation | 11 | 7
  Dilated with Tropicamide, 4 hr: Changed Accommodation (≥1 D) | 5 | 9
  Dilated with Phenylephrine, 0 min: number analyzed (Participants) | 15 | 15
  Dilated with Phenylephrine, 0 min: Unchanged Accommodation | 10 | 11
  Dilated with Phenylephrine, 0 min: Changed Accommodation (≥1 D) | 5 | 4
  Dilated with Phenylephrine, 2 hr: number analyzed (Participants) | 15 | 15
  Dilated with Phenylephrine, 2 hr: Unchanged Accommodation | 11 | 13
  Dilated with Phenylephrine, 2 hr: Changed Accommodation (≥1 D) | 4 | 2
  Dilated with Phenylephrine, 4 hr: number analyzed (Participants) | 15 | 15
  Dilated with Phenylephrine, 4 hr: Unchanged Accommodation | 12 | 13
  Dilated with Phenylephrine, 4 hr: Changed Accommodation (≥1 D) | 3 | 2

5. Secondary Outcome: Conjunctival Hyperemia (Eye Redness) Assessed Visually With the Brien Holden Vision Institute (Formerly Corneal and Contact Lens Research Unit, or CCLRU) Bulbar Redness Scale (0-3)
Description: Conjunctival hyperemia at each timepoint (0 min, 30 min, 1 hour, 2 hours, 4 hours, 6 hours), for study eye; in all subjects. Scale 0-3 (None, Mild, Moderate, Severe)
Time Frame: 0 min, 30 min, 1 hour, 2 hours, 4 hours, 6 hours
Population: All randomized participants who recieved the medication.
Measure: Mean (Standard Deviation); unit: score on a scale (0-3)
Arm/Group | Phentolamine Mesylate Ophthalmic Solution 1% | Phentolamine Mesylate Ophthalmic Solution Vehicle
Number analyzed (Participants) | 31 | 32
score on a scale (0-3)
  Baseline (-1 hr) | 0.45 (0.568) | 0.35 (0.486)
  0 min | 0.23 (0.497) | 0.29 (0.461)
  30 min | 1.52 (0.677) | 0.42 (0.502)
  1 hr | 1.55 (0.675) | 0.45 (0.568)
  2 hr | 1.42 (0.620) | 0.45 (0.568)
  4 hr | 1.10 (0.539) | 0.42 (0.564)
  6 hr | 0.81 (0.654) | 0.35 (0.486)

6. Secondary Outcome: Best Corrected Distance Visual Acuity (BCDVA) Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) Light Box Chart (Letters) at 4 Meters (Change From Baseline)
Description: Change from baseline (-1 hour) in Best Corrected Distance Visual Acuity at each time point (0 min, 30 mins, 1 hour, 2 hours, 6 hours) in Study Eye
Time Frame: 0 mins, 30 mins, 1 hour, 2 hours, 4 hours, 6 hours
Measure: Mean (Standard Error); unit: Letters Read
Arm/Group | Phentolamine Mesylate Ophthalmic Solution 1% | Phentolamine Mesylate Ophthalmic Solution Vehicle
Number analyzed (Participants) | 31 | 31
Letters Read
  0 mins | -0.45 (2.142) | -0.81 (2.182)
  30 mins | -0.55 (2.188) | -0.55 (1.690)
  1 hour | 0.29 (1.774) | -0.10 (2.797)
  2 hours | 0.65 (2.727) | 0.16 (2.162)
  4 hours | 1.06 (2.205) | 0.10 (2.119)
  6 hours | 0.45 (3.982) | 0.90 (2.399)

7. Secondary Outcome: Distance-Corrected Near Visual Acuity (DCNVA) Measured by Standard Reading Card (Original Series Sloan Letter ETDRS Card at 16 Inches, LogMAR Units) (Change From Baseline)
Description: Change from baseline (-1 hour) in Distance Corrected Near Visual Acuity at each time point (0 min, 30 mins, 1 hour, 2 hours, 6 hours) in Study Eye
Time Frame: 0 mins, 30 mins, 1 hour, 2 hours, 4 hours, 6 hours
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Phentolamine Mesylate Ophthalmic Solution 1% | Phentolamine Mesylate Ophthalmic Solution Vehicle
Number analyzed (Participants) | 31 | 31
LogMar
  0 mins | 0.14 (0.194) | 0.13 (0.216)
  30 mins | 0.09 (0.156) | 0.09 (0.217)
  1 hour | 0.05 (0.146) | 0.07 (0.142)
  2 hours | 0.03 (0.113) | 0.00 (0.087)
  4 hours | 0.00 (0.075) | 0.01 (0.079)
  6 hours | -0.02 (0.083) | 0.00 (0.055)

ADVERSE EVENTS:
Time Frame: 2 weeks.
Description: All AEs/adverse reactions occurring during the study (ie, once the subject had signed the informed consent) were documented on the CRF, regardless of the assumption of causal relationship. All TEAEs/adverse reactions were documented from the time the subject received the first dose of study medication until the subject's participation in the study had completed.
Arm/Group | Phentolamine Mesylate Ophthalmic Solution 1% | Phentolamine Mesylate Ophthalmic Solution Vehicle
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 11/31 | 1/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phentolamine Mesylate Ophthalmic Solution 1% (N=31) | Phentolamine Mesylate Ophthalmic Solution Vehicle (N=32)
Conjunctival Hyperemia (Eye disorders) | 11 | 0
Abdominal Pain, Upper (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT04024891/Prot_002.pdf
  • Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT04024891/SAP_003.pdf